CLINICAL TRIAL: NCT04738630
Title: A Single-arm, Open-lable, Multicenter, Phase II Clinical Study of HX008 in Subjects With BCG-Unresponsive Non-muscle Invasive Bladder Cancer
Brief Title: Study of HX008 for the Treatment of BCG-Unresponsive Non-muscle Invasive Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou Hanzhong biomedical co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX008-II-NMIBC-01
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: HX008 (Experimental): Participants will receive HX008 200 mg intravenous (IV) every 3 weeks (Q3W)
  Interventions: Drug: HX008

INTERVENTIONS:
Drug: HX008 — 200 mg administered as IV infusion on Day 1 of each 21-day cycle.

SUMMARY:
This is a single-arm, multicenter study to evaluate the efficacy and safety of HX008 injection in patients with BCG-unresponsive non-muscle invasive bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Age ≥ 18 years old, male or female.
* Predominant histologic component (> 50%) must be urothelial (transitional cell) carcinoma.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Score.
* Histologically-confirmed diagnosis of high risk non-muscle invasive bladder cancer (T1, high grade Ta and/or carcinoma in situ [CIS]).
* BCG-unresponsive high risk non-muscle-invasive bladder cancer, BCG-unresponsive disease as defined as: (a) Persistent or recurrent CIS (+/- recurrent Ta/T1 disease) within 9 months of receiving adequate BCG (at least five of six doses doses of an initial induction course plus either at least two of three doses of maintenance therapy or at least two of six doses of a second induction course); or (b) Recurrent high-grade Ta/T1 disease within 9 months of completion of adequate BCG (at least five of six doses of an initial induction course plus either at least two of three doses of maintenance therapy or at least two of six doses of a second induction course).
* Patients must be deemed unfit for radical cystectomy by the treating physician or refuse radical cystectomy.
* All visible tumor must be completely resected 60 days prior to the first dose of trial treatment. Patients with T1 tumors must undergo a re-staging transurethral resection of bladder tumor (TURBT) within 6 weeks after initial TURBT, and re-staging TURBT must be 60 days prior to the first dose of trial treatment.
* All patients must have had a cystoscopy without papillary tumor and negative urinary cytology within 21 days prior to the first dose of trial treatment (positive cytology is allowed in patients with CIS component). A cystoscopy is not needed if the TURBT falls within 21 days of prior to the first dose of trial treatment.
* Patients must have had imaging with X-ray for chest, computed tomography (CT) or magnetic resonance imaging (MRI) for abdomen/pelvis within 90 days prior to the first dose of trial treatment demonstrating no evidence of metastasis.
* Willing to provide tissue specimens.
* Has adequate organ function as defined in the protocol.
* Male subjects must agree to use effective contraceptives during treatment and for at least 120 days after the last treatment.
* Women of childbearing age must have a negative pregnancy test within 72 hours before the first dose of trial treatment, and agree to use effective contraceptives during treatment and for at least 120 days after the last treatment.

Exclusion Criteria:

* Muscle-invasive or metastatic urothelial carcinoma.
* Concurrent extra-vesical (i.e., urethra, ureter, or renal pelvis) non-muscle invasive transitional cell carcinoma of the urothelium.
* Patients who had a malignant tumor other than urothelial carcinoma of the bladder within the first 5 years of enrolment. The following can be included: a. low-risk localized prostate cancer (staging ≤ T2B, Gleason score ≤7, PSA≤20ng/mL, no recurrence after treatment (as determined by PSA level)); b. low-risk prostate cancer (T1/ T2A, Gleason score ≤7, and PSA≤10ng/mL) who were not treated and under observation; c. patients with very low risk metastasis or death of malignant tumor (5-year metastasis or death risk< 5%), showed no recurrence after standard treatment, such as cervical cancer in situ, basal or squamous cell skin cancer, etc.
* Has received prior therapy with an anti-PD-1, or anti-PD-L1, or anti-CTLA-4, or anti-4-1BB agents.
* Has received systemic chemotherapy or immunotherapy, or radiation therapy for bladder cancer.
* Patients with active autoimmune disease that has required systemic treatment in past 2 years.
* Has received a major surgery within 4 weeks prior to the first dose of trial treatment.
* Has a history of testing positive for human immunodeficiency virus (HIV), or known acquired immunodeficiency syndrome (AIDS), or stem cell transplantation or organ transplantation.
* Patients with active chronic hepatitis B or active hepatitis C. Patients with non-active HBsAg carriers, treated and stable hepatitis B (HBV DNA below the threshold of the test standard of each center), and cured hepatitis C can be enrolled.
* Has received system treatment with corticosteroids (dose >10mg/day prednison or other therapeutic hormones) within 2 weeks prior to the first dose of trial treatment.
* Has a history of active tuberculosis.
* Has a history or current interstitial pneumonia, or current non--infectious pneumonitis.
* Has uncontrolled systemic disease, such as diabetes or hypertension.
* Has cardiac dysfunction (grade III-IV according to NYHA) and significant pulmonary disease (such as shortness of breath at rest or minor activity or the need for oxygen for any reason) prior to the first dose of trial treatment.
* Patients with other disease, or metabolic disorder, or abnormal physical examination or laboratory test, or anticipated to cause complications with trial treatment.
* Has a severe infection prior to the first dose of trial treatment.
* Has a history of severe allergic reaction to any other monoclonal antibodies.
* Has participated in other anticancer drug clinical trials within 4 weeks.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | up to approximately 24 months
Event-free survival (EFS) | up to approximately 36 months

SECONDARY OUTCOMES:
Duration of response (DOR) | up to approximately 36 months
Event-free survival (EFS) in the Ta/T1 subset | up to approximately 36 months
Progression-free survival (PFS) | up to approximately 36 months
Recurrence free survival (RFS) | up to approximately 36 months
Overall survival (OS) | up to approximately 36 months
Cystectomy-free survival | up to approximately 36 months

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of science and technology, Wuhan, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of science and technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Sichuan